CLINICAL TRIAL: NCT03926728
Title: A Phase I, Double-blind, Parallel, Randomised and Placebo-controlled Trial Investigating the Safety and Immunogenicity of a Chlamydia Vaccine, CTH522, in Healthy Adults
Brief Title: Safety and Immunogenicity of a Chlamydia Vaccine CTH522
Acronym: CHLM-02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CHLM-02
Record Dates: First submitted 2019-04-15; First posted 2019-04-24 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-03

CONDITIONS: Trachoma
Keywords: CTH522; Chlamydia; C. Trachomatis
MeSH Terms: conditions — Trachoma; Chlamydia Infections | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort A 85 mcg CTH522-CAF01 (Experimental): Cohort A received three IM vaccination of 85 mcg CTH522-CAF01 (Day 0, 28, and 112). This cohort was divided into two groups: Cohort A1 receives placebo at Day 28, 112, and 140, while cohort A2 received placebo at Day 28 and 112, but non-adjuvanted TO CTH522 boost at Day 140.
  Interventions: Biological: CTH522-CAF01 IM; Biological: CTH522 TO; Biological: Placebo (Saline)
- Cohort B 85 mcg CTH522-CAF01 + TO CTH522 (Experimental): Cohort B received three IM vaccination of 85 mcg CTH522-CAF01 (Day 0, 28, and 112). This cohort was divided into two groups: Cohort B1 received TO vaccination of the non-adjuvanted CTH522 at Day 28 and 112 and TO placebo at Day 140, while cohort B2 received the same for Day 28 and 112, but non-adjuvanted TO CTH522 boost at Day 140.
  Interventions: Biological: CTH522-CAF01 IM; Biological: CTH522 TO; Biological: Placebo (Saline)
- Cohort C 85 mcg CTH522-CAF01 + ID CTH522 (Experimental): Cohort C received three IM vaccination of 85 mcg CTH522-CAF01 (Day 0, 28, and 112). This cohort was divided into two groups: Cohort C1 received ID vaccination of the non-adjuvanted CTH522 at Day 28 and 112 and TO placebo at Day 140, while cohort C2 received the same for Day 28 and 112, but TO CTH522 boost at Day 140.
  Interventions: Biological: CTH522-CAF01 IM; Biological: CTH522 ID; Biological: CTH522 TO; Biological: Placebo (Saline)
- Cohort D 15 mcg CTH522-CAF01 (Experimental): Cohort D received three IM vaccination of 15 mcg CTH522-CAF01 (Day 0, 28, and 112). This cohort was divided into two groups: Cohort D1 received TO placebo given on Day 28, 112, and 140, while cohort D2 received ID placebo given on Day 28 and 112 and TO unadjuvanted CTH522 on Day 140.
  Interventions: Biological: CTH522-CAF01 IM; Biological: CTH522 TO; Biological: Placebo (Saline)
- Cohort E 85 mcg CTH522-CAF09b (Experimental): Cohort E received three IM vaccination of 85 mcg CTH522-CAF09b (Day 0, 28, and 112). This cohort was divided into two groups: Cohort E1 received TO placebo given on Day 28, 112, and 140, while cohort E2 received ID placebo given on Day 28 and 112 and TO unadjuvanted CTH522 on Day 140.
  Interventions: Biological: CTH522-CAF09b IM; Biological: CTH522 TO; Biological: Placebo (Saline)
- Cohort F Placebo (Placebo Comparator): Cohort F received three IM vaccinations of placebo in form of 0.9% NaCl saline (Day 0, 28, and 112).This cohort was divided into two groups: Cohort F1 received TO placebo given on Day 28, 112, and 140, while cohort F2 received ID placebo given on Day 28 and 112 and TO placebo on Day 140.
  Interventions: Biological: Placebo (Saline)

INTERVENTIONS:
Biological: CTH522-CAF01 IM — On-site reconstitution of IMPs is performed by mixing 85 mcg CTH522 with CAF01. The preferred for IM is in the non-dominant deltoid muscle. IM injection will be performed with a 1-2 mL polypropylene Luer-Lok™ syringe via 23-25 gauge needle. The identity of the injected trial vaccine will be known to the clinical site staff dispensing and/or injecting the trial vaccine to the subject and by the unblinded trial monitor. The identity of the trial vaccine administered will remain unknown to the subject during the trial.
  Arms: Cohort A 85 mcg CTH522-CAF01; Cohort B 85 mcg CTH522-CAF01 + TO CTH522; Cohort C 85 mcg CTH522-CAF01 + ID CTH522; Cohort D 15 mcg CTH522-CAF01
Biological: CTH522-CAF09b IM — On-site reconstitution of IMPs is performed by mixing 85 mcg CTH522 with CAF09b. The preferred for IM is in the non-dominant deltoid muscle. IM injection will be performed with a 1-2 mL polypropylene Luer-Lok™ syringe via 23-25 gauge needle. The identity of the injected trial vaccine will be known to the clinical site staff dispensing and/or injecting the trial vaccine to the subject and by the unblinded trial monitor. The identity of the trial vaccine administered will remain unknown to the subject during the trial.
  Arms: Cohort E 85 mcg CTH522-CAF09b
Biological: CTH522 ID — 24 mcg CTH522 given ID is in the non-dominant deltoid muscle. ID with a 1 mL syringe via a 26-28 gauge needle using a NanoPass device or similar. The identity of the injected trial vaccine will be known to the clinical site staff dispensing and/or injecting the trial vaccine to the subject and by the unblinded trial monitor. The identity of the trial vaccine administered will remain unknown to the subject during the trial.
  Arms: Cohort C 85 mcg CTH522-CAF01 + ID CTH522
Biological: CTH522 TO — 24 mcg CTH522 (12 mcg in each eye) TO administrations will be performed using a Gilson positive displacement pipette. The identity of vaccine will be known to the clinical site staff dispensing/administrating the trial vaccine to the subject and by the unblinded trial monitor. The identity of the trial vaccine administered will remain unknown to the subject during the trial.
  Arms: Cohort A 85 mcg CTH522-CAF01; Cohort B 85 mcg CTH522-CAF01 + TO CTH522; Cohort C 85 mcg CTH522-CAF01 + ID CTH522; Cohort D 15 mcg CTH522-CAF01; Cohort E 85 mcg CTH522-CAF09b
Biological: Placebo (Saline) — Placebo only given as IM, ID and TO.

SUMMARY:
CHLM-02 was a phase I, double-blind, randomized, placebo-controlled trial of the chlamydia vaccine CTH522. 65 trial participants were randomized into 12 groups and six cohorts (A1 to F2). Cohorts A to E received three intramuscular (IM) injections of CTH522 (Day 0, 28, and 112). Cohorts A to D received CTH522 adjuvanted with Cationic Adjuvant Formulation (CAF®) 01 IM in two doses (85µg [A to C] or 15µg [D]). Cohort E received 85µg CTH522 adjuvanted with CAF®09b. Cohorts B and C received unadjuvanted CTH522 boost via the topic ocular (TO) or intradermal (ID) route, respectively, jointly with the second and third IM vaccinations. Cohort F received placebo. The effect of mucosal recall on eye immunity with TO CTH522 or placebo was assessed Day 140.

DETAILED DESCRIPTION:
This trial was a phase I, double-blind, parallel, randomised, and placebo-controlled trial of the chlamydia vaccine CTH522 in healthy adults.

It was planned to randomize 66 subjects but only 65 subjects were randomized. Cohorts A-D investigated CTH522-CAF01 administered IM in two doses (85 mcg and 15 mcg). Cohort E investigated CTH522-CAF09b administered IM in one dose (85 mcg). Cohort F was the placebo group. The enrolled subjects were to complete 12 trial visits. All subjects in the active cohorts (cohort A-E) were to receive three IM injections of the adjuvanted CTH522 and some (cohort B and C) were to receive the non-adjuvanted CTH522 via the TO or ID route (given at the same time as the 2nd and 3rd IM vaccinations). All active cohorts were to receive TO administration as a boost at Day 140 of either the non-adjuvanted CTH522 (12 mcg in each eye) or placebo.

* Cohort A received three IM vaccination of 85 mcg CTH522-CAF01. This cohort was divided into two groups: A1 received ID placebo at Day 28 and Day 112, and TO placebo at Day 140, while A2 received TO placebo at Day 28 and Day 112, and non-adjuvanted TO CTH522 boost at Day 140.
* Cohort B received three IM vaccinations of 85 mcg CTH522-CAF01. This cohort was divided into two groups: B1 received TO vaccination of the non-adjuvanted CTH522 at Day 28 and 112 and TO placebo at Day 140, while B2 received the same for Day 28 and 112, but non-adjuvanted TO CTH522 boost at Day 140. The two additional TO doses of CTH522 (12 mcg in each eye) were administered in each eye. The rationale for this schedule was to investigate the impact of simultaneous TO administration of the antigen on the immunogenicity results.
* Cohort C received three IM vaccinations of 85 mcg CTH522-CAF01. This cohort was divided into two groups: C1 received ID vaccination of the non-adjuvanted 24 mcg CTH522 at Day 28 and 112 and TO placebo at Day 140, while C2 received the same for Day 28 and 112, but TO 12 mcg CTH522 boost in each eye at Day 140. The rationale for this schedule was to investigate the impact of simultaneous ID administration of the antigen on the immunogenicity results.
* Cohort D received three IM vaccinations of 15 mcg CTH522-CAF01. The rationale for the A and D cohorts was to investigate the impact of the two IM CTH522 doses on the immunogenicity results.
* Cohort E received three IM vaccinations of 85 mcg CTH522-CAF09b. The rationale for the A and E cohorts was to investigate the impact of the adjuvant on the immunogenicity results.
* Cohort F received placebo in the form of 0.9% NaCl saline (IM, ID and TO).

ELIGIBILITY:
Inclusion Criteria:

IC1: Healthy males and females between 18-45 years old on the day of the first vaccination.

IC2: Has been properly informed about the trial and signed the consent form.

IC3: Is willing and likely to comply with trial procedures.

IC4: Is prepared to grant authorised persons access to his/her trial-related medical record.

IC5: Is willing to use acceptable contraceptive measures during the trial (two weeks before and two weeks after the trial). Heterosexually active female capable of becoming pregnant must agree to use hormonal contraception, intrauterine device, intrauterine hormone releasing system, or to complete abstinence from at least two weeks before the first vaccination until at least two weeks after the last. Complete abstinence (defined as refraining from heterosexual intercourse) must be in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods), withdrawal and progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action, are not acceptable methods of contraception.

Exclusion criteria:

EX1: Is positive for C. trachomatis via urine PCR or has a known history of C. trachomatis.

EX2: Is positive for gonorrhoea via urine PCR test, or HIV, hepatitis B/C, syphilis via blood tests.

EX3: Has a significant active disease such as cardiac, liver, immunological, neurological, psychiatric, or clinically significant abnormality of haematological or biochemical parameters.

EX4: Has BMI ≥ 35 kg/m2.

EX5: Is currently participating in another clinical trial with an investigational or noninvestigational drug or device, or was treated with an investigational drug within 28 days before the first vaccination.

EX6: Has received, or plans to receive, any immunisation within 14 days of the start of the trial or during the trial immunisations.

EX7: Is currently receiving treatment with systemic immunosuppressive agents. Topical steroids are allowed unless applied to the IM or ID injection site.

EX8: Has a condition which in the opinion of the investigator is not suitable for participation in the trial.

EX9: Is known or confirmed to have an allergy to any of the vaccine constituents.

EX10: Is unable to refrain from the use of contact lenses. Contact lenses should be avoided two days before TO administration and for seven days later (longer if any ongoing local eye AE).

EX11: Has any evident ocular disease upon ophthalmoscopic exam at screening or any medical history of ocular disease that, in the opinion of the investigator, may impact the subject's participation in the trial.

EX12: Is pregnant (positive pregnancy test) or breastfeeding or not willing to use contraception during the trial.

EX13: Has confirmed a history of pelvic inflammatory disease or significant gynaecological diseases.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Borges, MD, Study Director — Statens Serum Institut; Katrina Pollock, MD, Principal Investigator — Imperial Clinical Research Facility Hammersmith Hospital; Lina S Stoey, MPH, Study Chair — Statens Serum Institut; Pernille N Tingskov, BS, Study Chair — Statens Serum Institut; Rebecca B Dohn, Pharm, Study Chair — Statens Serum Institut
Locations (1):
- NIHR Imperial Center for Translational and Experimental Medicine, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pollock KM, Borges AH, Cheeseman HM, Rosenkrands I, Schmidt KL, Sondergaard RE, Day S, Evans A, McFarlane LR, Joypooranachandran J, Amini F, Skallerup P, Dohn RB, Jensen CG, Olsen AW, Bang P, Cole T, Schronce J, Lemm NM, Kristiansen MP, Andersen PL, Dietrich J, Shattock RJ, Follmann F. An investigation of trachoma vaccine regimens by the chlamydia vaccine CTH522 administered with cationic liposomes in healthy adults (CHLM-02): a phase 1, double-blind trial. Lancet Infect Dis. 2024 Aug;24(8):829-844. doi: 10.1016/S1473-3099(24)00147-6. Epub 2024 Apr 11. PMID 38615673

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo: Participants received 3 IM vaccinations of 85 mcg CTH522-CAF01 (Day 0, 28, and 112). In addition, participants received ID placebo given on Day 28 and 112 and TO placebo given on Day 140.
- Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522: Participants received 3 IM vaccinations of 85 mcg CTH522-CAF01 (Day 0, 28, and 112). In addition, participants received TO placebo given on Day 28 and 112 and TO unadjuvanted CTH522 given on Day 140.
- Cohort B1 85 mcg IM CTH522-CAF01+ TO CTH522 + TO Placebo: Participants received 3 IM vaccinations of 85 mcg CTH522-CAF01 (Day 0, 28, and 112). In addition, participants received TO unadjuvanted CTH522 given on Day 28 and 112 and TO placebo given on Day 140.
- Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522: Participants received 3 IM vaccinations of 85 mcg CTH522-CAF01 (Day 0, 28, and 112). In addition, participants received TO unadjuvanted CTH522 given on Day 28, 112, and 140.
- Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo: Participants received 3 IM vaccinations of 85 mcg CTH522-CAF01 (Day 0, 28, and 112). In addition, participants received ID unadjuvanted CTH522 given on Day 28 and 112 and TO placebo given on Day 140.
- Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522: Participants received 3 IM vaccinations of 85 mcg CTH522-CAF01 (Day 0, 28, and 112). In addition, participants received ID unadjuvanted CTH522 given on Day 28 and 112 and TO unadjuvanted CTH522 given on Day 140.
- Cohort D1 15 mcg IM CTH522-CAF01 + TO Placebo: Participants received 3 IM vaccinations of 15 mcg CTH522-CAF01 (Day 0, 28, and 112). In addition, participants received TO placebo given on Day 28, 112, and 140.
- Cohort D2 15 mcg IM CTH522-CAF01 + ID Placebo + TO CTH522: Participants received 3 IM vaccinations of 15 mcg CTH522-CAF01 (Day 0, 28, and 112). In addition, participants received ID placebo given on Day 28 and 112 and TO unadjuvanted CTH522 on Day 140.
- Cohort E1 85 mcg IM CTH522-CAF09b + TO Placebo: Participants received 3 IM vaccinations of 85 mcg CTH522-CAF09b (Day 0, 28, and 112). In addition, participants received TO placebo given on Day 28, 112, and 140.
- Cohort E2 85 mcg IM CTH522-CAF09b + ID Placebo + TO CTH522: Participants received 3 IM vaccinations of 85 mcg CTH522-CAF09b (Day 0, 28, and 112). In addition, participants received ID placebo given on Day 28 and 112 and TO unadjuvanted CTH522 on Day 140.
- Cohort F1 IM Placebo + TO Placebo: Participants received 3 IM vaccinations of placebo (Day 0, 28, and 112). In addition, participants received TO placebo given on Day 28, 112, and 140.
- Cohort F2 IM Placebo + ID Placebo + TO Placebo: Participants received 3 IM vaccinations of placebo (Day 0, 28, and 112). In addition, participants received ID placebo given on Day 28 and 112 and TO placebo on Day 140.
Period: Overall Study
Arm/Group | Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo | Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 | Cohort B1 85 mcg IM CTH522-CAF01+ TO CTH522 + TO Placebo | Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 | Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo | Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 | Cohort D1 15 mcg IM CTH522-CAF01 + TO Placebo | Cohort D2 15 mcg IM CTH522-CAF01 + ID Placebo + TO CTH522 | Cohort E1 85 mcg IM CTH522-CAF09b + TO Placebo | Cohort E2 85 mcg IM CTH522-CAF09b + ID Placebo + TO CTH522 | Cohort F1 IM Placebo + TO Placebo | Cohort F2 IM Placebo + ID Placebo + TO Placebo
Started | 2 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 3
Completed | 2 | 8 | 2 | 9 | 3 | 8 | 2 | 9 | 3 | 8 | 3 | 3
Not Completed | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo: Participants received 3 IM vaccinations of 85 mcg CTH522-CAF01 (Day 0, 28, and 112). In addition, participants received TO unadjuvanted CTH522 given on Day 28 and 112 and TO placebo given on Day 140.
- Total: Total of all reporting groups
Arm/Group | Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo | Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 | Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo | Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 | Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo | Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 | Cohort D1 15 mcg IM CTH522-CAF01 + TO Placebo | Cohort D2 15 mcg IM CTH522-CAF01 + ID Placebo + TO CTH522 | Cohort E1 85 mcg IM CTH522-CAF09b + TO Placebo | Cohort E2 85 mcg IM CTH522-CAF09b + ID Placebo + TO CTH522 | Cohort F1 IM Placebo + TO Placebo | Cohort F2 IM Placebo + ID Placebo + TO Placebo | Total
Number analyzed (Participants) | 2 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 3 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 3 | 65
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.0 (1.4) | 26.9 (6.4) | 21.7 (2.1) | 28.4 (7.3) | 32.3 (6.1) | 22.4 (2.4) | 25.7 (9) | 26.8 (5.6) | 31.7 (8.5) | 30.1 (9.9) | 24.7 (5.5) | 25.0 (5.3) | 26.8 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 5 | 1 | 1 | 1 | 6 | 2 | 5 | 3 | 5 | 2 | 3 | 34
  Male | 2 | 4 | 2 | 8 | 2 | 3 | 1 | 4 | 0 | 4 | 1 | 0 | 31
Race/Ethnicity, Customized [Number; unit: participants]
  White | 1 | 6 | 3 | 4 | 3 | 6 | 3 | 6 | 1 | 7 | 3 | 3 | 46
  Asian | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 1 | 1 | 1 | 0 | 0 | 8
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3
  Other | 1 | 1 | 0 | 4 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 8
Region of Enrollment [Number; unit: participants]
  United Kingdom | 2 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 3 | 65
BMI [Mean (Standard Deviation); unit: kg/m2] | 20.70 (3.96) | 24.78 (3.02) | 23.73 (2.25) | 22.62 (3.58) | 26.23 (2.55) | 23.63 (2.41) | 24.70 (1.55) | 23.13 (1.67) | 21.70 (0.92) | 24.11 (3.55) | 24.37 (3.20) | 22.77 (0.55) | 23.64 (2.78)

OUTCOME MEASURES:

1. Primary Outcome: Solicited Local Injection Site Reactions
Description: Local injection site reactions after intramuscular vaccination. Solicited local injection site reactions are defined as erythema, pruritus, pain, tenderness, swelling, and warmth.
Time Frame: Visit 2 (Day 0) plus 14 Days
Measure: Count of Participants; unit: Participants
Groups:
- Cohort D1 15 mcg IM CTH522-CAF01 + TO Placebo: Participants received 3 IM vaccinations of 15 mcg CTH522-CAF01 (Day 0, 28, and 112). In addition, participants received TO placebo given on Day 28,112, and 140.
- Cohort E1 85 mcg IM CTH522-CAF09b + TO Placebo: Participants received 3 IM vaccinations of 85 mcg CTH522-CAF09b (Day 0, 28, and 112). In addition, participants received TO placebo given on Day 28,112, and 140.
- Cohort F2 IM Placebo + ID Placebo + TO Placebo: Participants received 3 IM vaccinations of placebo (Day 0, 28 ,and 112). In addition, participants received ID placebo given on Day 28 and 112 and TO placebo on Day 140.
Arm/Group | Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo | Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 | Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo | Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 | Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo | Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 | Cohort D1 15 mcg IM CTH522-CAF01 + TO Placebo | Cohort D2 15 mcg IM CTH522-CAF01 + ID Placebo + TO CTH522 | Cohort E1 85 mcg IM CTH522-CAF09b + TO Placebo | Cohort E2 85 mcg IM CTH522-CAF09b + ID Placebo + TO CTH522 | Cohort F1 IM Placebo + TO Placebo | Cohort F2 IM Placebo + ID Placebo + TO Placebo
Number analyzed (Participants) | 2 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 3
Participants
  Injection site pain | 2 | 8 | 3 | 9 | 2 | 9 | 3 | 9 | 3 | 9 | 0 | 1
  Injection site warmth | 0 | 1 | 2 | 3 | 1 | 4 | 0 | 2 | 1 | 2 | 0 | 1
  Injection site swelling | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0
  Injection site erythema | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
  Injection site pruritus | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Statistical Analysis 1: Comparison: Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo vs Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 vs Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo vs Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 vs Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo vs Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 vs Cohort D1 15 mcg IM CTH522-CAF01 + TO Placebo vs Cohort D2 15 mcg IM CTH522-CAF01 + ID Placebo + TO CTH522; Comparison: Cohort A-C [A1, A2, B1, B2, C1, C2] vs D [D1, D2]; Test type: Other; p = 1, Fisher Exact — Simple nonparametric statistical test
Statistical Analysis 2: Comparison: Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo vs Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 vs Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo vs Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 vs Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo vs Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 vs Cohort E1 85 mcg IM CTH522-CAF09b + TO Placebo vs Cohort E2 85 mcg IM CTH522-CAF09b + ID Placebo + TO CTH522; Comparison: Cohort A-C [A1, A2, B1, B2, C1, C2] vs E [E1, E2]; Test type: Other; p = 1, Fisher Exact — Simple nonparametric statistical test
Statistical Analysis 3: Comparison: Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo vs Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 vs Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo vs Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 vs Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo vs Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 vs Cohort F1 IM Placebo + TO Placebo vs Cohort F2 IM Placebo + ID Placebo + TO Placebo; Comparison: Cohort A-C [A1, A2, B1, B2, C1, C2] vs F [F1, F2]; Test type: Other; p = 0.0007, Fisher Exact

2. Primary Outcome: Solicited Local Injection Site Reactions
Description: Local injection site reactions after intramuscular vaccination (participants also received intradermal or topical ocular administration of CTH522 or placebo). Solicited local injection site reactions are defined as erythema, pruritus, pain, tenderness, swelling, and warmth.
Time Frame: Visit 4 (Day 28) plus 14 Days
Population: Percentages calculated from number of participants vaccinated on Day 28.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo | Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 | Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo | Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 | Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo | Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 | Cohort D1 15 mcg IM CTH522-CAF01 + TO Placebo | Cohort D2 15 mcg IM CTH522-CAF01 + ID Placebo + TO CTH522 | Cohort E1 85 mcg IM CTH522-CAF09b + TO Placebo | Cohort E2 85 mcg IM CTH522-CAF09b + ID Placebo + TO CTH522 | Cohort F1 IM Placebo + TO Placebo | Cohort F2 IM Placebo + ID Placebo + TO Placebo
Number analyzed (Participants) | 2 | 9 | 2 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 3
Participants
  Injection site pain | 2 | 8 | 2 | 9 | 3 | 9 | 2 | 9 | 3 | 6 | 1 | 2
  Injection site warmth | 0 | 3 | 1 | 3 | 0 | 2 | 0 | 2 | 0 | 1 | 1 | 1
  Injection site erythema | 0 | 0 | 0 | 0 | 3 | 4 | 0 | 0 | 0 | 2 | 0 | 1
  Injection site pruritus | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 0
  Injection site swelling | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 0 | 1

3. Primary Outcome: Solicited Local Injection Site Reactions
Description: as for outcome 2
Time Frame: Visit 7 (Day 112) plus 14 Days
Population: Percentages calculated from number of participants vaccinated on Day 112
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo | Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 | Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo | Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 | Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo | Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 | Cohort D1 15 mcg IM CTH522-CAF01 + TO Placebo | Cohort D2 15 mcg IM CTH522-CAF01 + ID Placebo + TO CTH522 | Cohort E1 85 mcg IM CTH522-CAF09b + TO Placebo | Cohort E2 85 mcg IM CTH522-CAF09b + ID Placebo + TO CTH522 | Cohort F1 IM Placebo + TO Placebo | Cohort F2 IM Placebo + ID Placebo + TO Placebo
Number analyzed (Participants) | 2 | 8 | 2 | 9 | 3 | 9 | 2 | 9 | 3 | 8 | 3 | 3
Participants
  Injection site pain | 1 | 6 | 2 | 8 | 2 | 8 | 1 | 7 | 2 | 8 | 2 | 0
  Injection site erythema | 0 | 0 | 0 | 2 | 3 | 6 | 0 | 1 | 1 | 3 | 1 | 0
  Injection site warmth | 0 | 2 | 1 | 1 | 1 | 5 | 0 | 2 | 0 | 3 | 1 | 1
  Injection site swelling | 0 | 1 | 1 | 0 | 2 | 3 | 1 | 1 | 0 | 3 | 0 | 0
  Injection site pruritus | 0 | 1 | 0 | 2 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 0

4. Primary Outcome: Solicited Local Ocular Reactions
Description: Local ocular reactions after topical ocular administration of CTH522 or placebo. Solicited local ocular reactions are defined as watering eyes, swelling of eyelid, eye redness, and eye discomfort.
Time Frame: Visit 4 (Day 28) plus 14 Days
Population: Percentages calculated from number of participants vaccinated on Day 28
Measure: Count of Participants; unit: Participants
Groups:
- Cohort F1 IM Placebo + TO Placebo: Participants received 3 IMvaccinations of placebo (Day 0, 28, and 112). In addition, participants received TO placebo given on Day 28, 112, and 140.
- Cohort F2 IM Placebo + ID Placebo + TO Placebo: Participants received 3 IMvaccinations of placebo (Day 0, 28, and 112). In addition, participants received ID placebo given on Day 28 and 112 and TO placebo on Day 140.
Arm/Group | Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo | Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 | Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo | Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 | Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo | Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 | Cohort D1 15 mcg IM CTH522-CAF01 + TO Placebo | Cohort D2 15 mcg IM CTH522-CAF01 + ID Placebo + TO CTH522 | Cohort E1 85 mcg IM CTH522-CAF09b + TO Placebo | Cohort E2 85 mcg IM CTH522-CAF09b + ID Placebo + TO CTH522 | Cohort F1 IM Placebo + TO Placebo | Cohort F2 IM Placebo + ID Placebo + TO Placebo
Number analyzed (Participants) | 2 | 9 | 2 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 3
Participants
  Ocular discomfort | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
  Lacrimation increased | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  Ocular hyperaemia | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Swelling of eyelid | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 vs Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo vs Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522; Comparison: Cohort B [B1, B2] vs A2; Test type: Other; p = 1, Fisher Exact — Simple nonparametric statistical test
Statistical Analysis 2: Comparison: Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo vs Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 vs Cohort F1 IM Placebo + TO Placebo; Comparison: Cohort B [B1, B2] vs F1; Test type: Other; p = 0.3956, Fisher Exact

5. Primary Outcome: Solicited Local Ocular Reactions
Description: as for outcome 4
Time Frame: Visit 7 (Day 112) plus 14 Days
Population: Percentages calculated from number of participants vaccinated on Day 112
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo: Participants received 3 IM vaccinations of 85 mcg CTH522-CAF01 (Day0, 28, and 112). In addition, participants received ID placebo given on Day 28 and112 and TO placebo given on Day 140.
- Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522: Participants received 3 IM vaccinations of 85 mcg CTH522-CAF01 (Day 0, 28, and 112). In addition, participants received TO placebo given on Day 28 and 112 and TO unadjuvanted CTH522 given on Day140.
- Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo: Participants received 3 IM vaccinations of 85 mcg CTH522-CAF01 (Day 0, 28, and 112). In addition, participants received TO unadjuvanted CTH522 given on Day 28 and 112 and TO placebo given on Day140.
- Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522: Participants received 3 IM vaccinations of 85 mcg CTH522-CAF01 (Day 0, 28, and 112). In addition, participants received ID unadjuvanted CTH522 given on Day 28 and 112 and TO unadjuvanted CTH522 given on Day140.
Arm/Group | Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo | Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 | Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo | Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 | Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo | Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 | Cohort D1 15 mcg IM CTH522-CAF01 + TO Placebo | Cohort D2 15 mcg IM CTH522-CAF01 + ID Placebo + TO CTH522 | Cohort E1 85 mcg IM CTH522-CAF09b + TO Placebo | Cohort E2 85 mcg IM CTH522-CAF09b + ID Placebo + TO CTH522 | Cohort F1 IM Placebo + TO Placebo | Cohort F2 IM Placebo + ID Placebo + TO Placebo
Number analyzed (Participants) | 2 | 8 | 2 | 9 | 3 | 9 | 2 | 9 | 3 | 8 | 3 | 3
Participants
  Ocular discomfort | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Ocular hyperaemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Lacrimation increased | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 vs Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo vs Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522; Comparison: Cohort B [B1, B2] vs A2; Test type: Other; p = 1, Fisher Exact — Simple nonparametric statistical test
Statistical Analysis 2: Comparison: Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo vs Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 vs Cohort F1 IM Placebo + TO Placebo; Comparison: Cohort B [B1, B2] vs F1; Test type: Other; p = 0.3956, Fisher Exact

6. Primary Outcome: Solicited Local Ocular Reactions
Description: as for outcome 4
Time Frame: Visit 9 (Day 140) plus 14 Days
Population: Percentages calculated from number of participants vaccinated on Day 140
Measure: Count of Participants; unit: Participants
Groups:
- Cohort F IM Placebo + TO Placebo: Participants received 3 IM vaccinations of placebo (Day 0, 28, and 112). In addition, participants received either TO placebo or ID placebo given on Day 28 and 112 and TO placebo given on Day 140.
Arm/Group | Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo | Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 | Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo | Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 | Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo | Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 | Cohort D1 15 mcg IM CTH522-CAF01 + TO Placebo | Cohort D2 15 mcg IM CTH522-CAF01 + ID Placebo + TO CTH522 | Cohort E1 85 mcg IM CTH522-CAF09b + TO Placebo | Cohort E2 85 mcg IM CTH522-CAF09b + ID Placebo + TO CTH522 | Cohort F IM Placebo + TO Placebo | Cohort F2 IM Placebo + ID Placebo + TO Placebo
Number analyzed (Participants) | 2 | 7 | 2 | 9 | 3 | 8 | 2 | 9 | 3 | 8 | 3 | 3
Participants
  Ocular discomfort | 0 | 2 | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 3 | 1 | 0
  Lacrimation increased | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
  Ocular hyperaemia | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 2 | 1 | 0
  Swelling of eyelid | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0

7. Primary Outcome: Solicited Systemic Reactions
Description: Systemic reactions after vaccinations. Solicited systemic reactions are defined as oral temperature > 38.3°C, chills, myalgia, and rash.
Time Frame: Visit 2 (Day 0) plus 14 Days
Population: Percentages calculated from number of participants vaccinated on Day 0
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo: Participants received 3 IM vaccinations of 85 mcg CTH522-CAF01 (Day 0, 28, and 112). In addition, participants received ID placebo given on Day 28 and 112 and TO placebogiven on Day 140.
Arm/Group | Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo | Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 | Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo | Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 | Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo | Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 | Cohort D1 15 mcg IM CTH522-CAF01 + TO Placebo | Cohort D2 15 mcg IM CTH522-CAF01 + ID Placebo + TO CTH522 | Cohort E1 85 mcg IM CTH522-CAF09b + TO Placebo | Cohort E2 85 mcg IM CTH522-CAF09b + ID Placebo + TO CTH522 | Cohort F1 IM Placebo + TO Placebo | Cohort F2 IM Placebo + ID Placebo + TO Placebo
Number analyzed (Participants) | 2 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 3
Participants
  Myalgia | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 2 | 0 | 0 | 0
  Chills | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Pyrexia | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo vs Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 vs Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo vs Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 vs Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo vs Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 vs Cohort D1 15 mcg IM CTH522-CAF01 + TO Placebo vs Cohort D2 15 mcg IM CTH522-CAF01 + ID Placebo + TO CTH522; Comparison: Cohort A-C [A1, A2, B1, B2, C1, C2] vs D [D1, D2]; Test type: Other; p = 1, Fisher Exact — Simple nonparametric statistical test
Statistical Analysis 2: Comparison: Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo vs Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 vs Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo vs Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 vs Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo vs Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 vs Cohort E1 85 mcg IM CTH522-CAF09b + TO Placebo vs Cohort E2 85 mcg IM CTH522-CAF09b + ID Placebo + TO CTH522; Comparison: Cohort A-C [A1, A2, B1, B2, C1, C2] vs E [E1, E2]; Test type: Other; p = 1, Fisher Exact — Simple nonparametric statistical test
Statistical Analysis 3: Comparison: Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo vs Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 vs Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo vs Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 vs Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo vs Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 vs Cohort F1 IM Placebo + TO Placebo vs Cohort F2 IM Placebo + ID Placebo + TO Placebo; Comparison: Cohort A-C [A1, A2, B1, B2, C1, C2] vs F [F1, F2]; Test type: Other; p = 0.3229, Fisher Exact

8. Primary Outcome: Solicited Systemic Reactions
Description: as for outcome 7
Time Frame: Visit 4 (Day 28) plus 14 Days
Population: Percentages calculated from number of participants vaccinated on Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo | Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 | Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo | Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 | Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo | Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 | Cohort D1 15 mcg IM CTH522-CAF01 + TO Placebo | Cohort D2 15 mcg IM CTH522-CAF01 + ID Placebo + TO CTH522 | Cohort E1 85 mcg IM CTH522-CAF09b + TO Placebo | Cohort E2 85 mcg IM CTH522-CAF09b + ID Placebo + TO CTH522 | Cohort F1 IM Placebo + TO Placebo | Cohort F2 IM Placebo + ID Placebo + TO Placebo
Number analyzed (Participants) | 2 | 9 | 2 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 3
Participants
  Myalgia | 0 | 3 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Chills | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0
  Rash | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Pyrexia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Solicited Systemic Reactions
Description: as for outcome 7
Time Frame: Visit 7 (Day 112) plus 14 Days
Population: Percentages calculated from number of participants vaccinated on Day 112
Measure: Count of Participants; unit: Participants
Groups:
- Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522: Participants received 3 IM vaccinations of 85 mcg CTH522-CAF01 (Day0, 28, and 112). In addition, participants received TO placebo given on Day 28 and 112 and TO unadjuvanted CTH522 given on Day 140.
- Cohort D2 15 mcg IM CTH522-CAF01 + ID Placebo + TO CTH522: Participants received 3 IM vaccinationsof 15 mcg CTH522-CAF01 (Day 0, 28, and 112). In addition, participants received ID placebo given on Day 28 and 112 and TO unadjuvanted CTH522 on Day 140.
- Cohort E1 85 mcg IM CTH522-CAF09b + TO Placebo: Participants received 3 IM vaccinations of 85 mcg CTH522-CAF09b (Day 0, 28, and 112). In addition, participants received TO placebogiven on Day 28, 112, and 140.
Arm/Group | Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo | Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 | Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo | Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 | Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo | Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 | Cohort D1 15 mcg IM CTH522-CAF01 + TO Placebo | Cohort D2 15 mcg IM CTH522-CAF01 + ID Placebo + TO CTH522 | Cohort E1 85 mcg IM CTH522-CAF09b + TO Placebo | Cohort E2 85 mcg IM CTH522-CAF09b + ID Placebo + TO CTH522 | Cohort F1 IM Placebo + TO Placebo | Cohort F2 IM Placebo + ID Placebo + TO Placebo
Number analyzed (Participants) | 2 | 8 | 2 | 9 | 3 | 9 | 2 | 9 | 3 | 8 | 3 | 3
Participants
  Myalgia | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 0 | 0
  chills | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 2 | 0 | 0

10. Secondary Outcome: Immunogenicity (4-fold Increase From Baseline)
Description: Frequency of 4-fold increase seroconversion from baseline for anti-CTH522 IgG after vaccinations.
Time Frame: Day 14, 28, 42, 56, 112, 126, 140, 154, 238
Population: Frequency of 4-fold increase seroconversion for anti-CTH522 IgG - full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo | Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 | Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo | Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 | Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo | Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 | Cohort D1 15 mcg IM CTH522-CAF01 + TO Placebo | Cohort D2 15 mcg IM CTH522-CAF01 + ID Placebo + TO CTH522 | Cohort E1 85 mcg IM CTH522-CAF09b + TO Placebo | Cohort E2 85 mcg IM CTH522-CAF09b + ID Placebo + TO CTH522 | Cohort F1 IM Placebo + TO Placebo | Cohort F2 IM Placebo + ID Placebo + TO Placebo
Number analyzed (Participants) | 2 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 3
Participants
  Day 14 | 0 | 6 | 2 | 7 | 2 | 7 | 1 | 2 | 3 | 7 | 0 | 0
  Day 28 | 0 | 8 | 1 | 6 | 2 | 6 | 2 | 2 | 3 | 6 | 0 | 0
  Day 42 | 2 | 8 | 2 | 9 | 3 | 9 | 3 | 9 | 3 | 8 | 0 | 0
  Day 56 | 2 | 8 | 2 | 9 | 3 | 8 | 3 | 9 | 3 | 8 | 0 | 0
  Day 112 | 1 | 8 | 2 | 9 | 3 | 9 | 2 | 9 | 3 | 8 | 0 | 0
  Day 126 | 2 | 8 | 2 | 9 | 3 | 8 | 2 | 9 | 3 | 8 | 0 | 0
  Day 140 | 2 | 8 | 2 | 9 | 3 | 8 | 2 | 9 | 3 | 8 | 0 | 0
  Day 154 | 2 | 8 | 2 | 9 | 3 | 8 | 2 | 9 | 3 | 8 | 0 | 0
  Day 238 | 2 | 8 | 2 | 9 | 3 | 7 | 2 | 9 | 3 | 8 | 0 | 0

11. Secondary Outcome: Immunogenicity (10-fold Increase From Baseline)
Description: Frequency of 10-fold increase seroconversion from baseline for anti-CTH522 IgG after vaccinations.
Time Frame: Day 14, 28, 42, 56, 112, 126, 140, 154, 238
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo | Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 | Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo | Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 | Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo | Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 | Cohort D1 15 mcg IM CTH522-CAF01 + TO Placebo | Cohort D2 15 mcg IM CTH522-CAF01 + ID Placebo + TO CTH522 | Cohort E1 85 mcg IM CTH522-CAF09b + TO Placebo | Cohort E2 85 mcg IM CTH522-CAF09b + ID Placebo + TO CTH522 | Cohort F1 IM Placebo + TO Placebo | Cohort F2 IM Placebo + ID Placebo + TO Placebo
Number analyzed (Participants) | 2 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 9 | 3 | 3
Participants
  Day 14 | 0 | 5 | 1 | 5 | 2 | 3 | 0 | 0 | 3 | 6 | 0 | 0
  Day 28 | 0 | 5 | 1 | 5 | 2 | 4 | 1 | 1 | 3 | 6 | 0 | 0
  Day 42 | 1 | 8 | 2 | 9 | 3 | 9 | 3 | 8 | 3 | 8 | 0 | 0
  Day 56 | 1 | 8 | 2 | 9 | 3 | 8 | 3 | 9 | 3 | 8 | 0 | 0
  Day 112 | 1 | 8 | 2 | 9 | 3 | 9 | 2 | 8 | 3 | 8 | 0 | 0
  Day 126 | 2 | 8 | 2 | 9 | 3 | 8 | 2 | 9 | 3 | 8 | 0 | 0
  Day 140 | 2 | 8 | 2 | 9 | 3 | 8 | 2 | 9 | 3 | 8 | 0 | 0
  Day 154 | 2 | 8 | 2 | 9 | 3 | 8 | 2 | 9 | 3 | 8 | 0 | 0
  Day 238 | 1 | 8 | 2 | 9 | 3 | 7 | 2 | 8 | 3 | 8 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 238 days after first vaccination
Description: The safety analysis set included all subjects who were randomised and exposed to at least one dosage of the study vaccine including subjects who were withdrawn after exposure to the study vaccine.
Arm/Group | Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo | Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 | Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo | Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 | Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo | Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 | Cohort D1 15 mcg IM CTH522-CAF01 + TO Placebo | Cohort D2 15 mcg IM CTH522-CAF01 + ID Placebo + TO CTH522 | Cohort E1 85 mcg IM CTH522-CAF09b + TO Placebo | Cohort E2 85 mcg IM CTH522-CAF09b + ID Placebo + TO CTH522 | Cohort F1 IM Placebo + TO Placebo | Cohort F2 IM Placebo + ID Placebo + TO Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/9 | 0/3 | 0/9 | 0/3 | 0/9 | 0/3 | 0/9 | 0/3 | 0/9 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/9 | 0/3 | 0/9 | 0/3 | 0/9 | 0/3 | 0/9 | 0/3 | 0/9 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 9/9 | 3/3 | 9/9 | 3/3 | 9/9 | 3/3 | 9/9 | 3/3 | 9/9 | 3/3 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A1 85 mcg IM CTH522-CAF01 + ID Placebo + TO Placebo (N=2) | Cohort A2 85 mcg IM CTH522-CAF01 + TO Placebo + TO CTH522 (N=9) | Cohort B1 85 mcg IM CTH522-CAF01 + TO CTH522 + TO Placebo (N=3) | Cohort B2 85 mcg IM CTH522-CAF01 + TO CTH522 (N=9) | Cohort C1 85 mcg IM CTH522-CAF01 + ID CTH522 + TO Placebo (N=3) | Cohort C2 85 mcg IM CTH522-CAF01 + ID CTH522 + TO CTH522 (N=9) | Cohort D1 15 mcg IM CTH522-CAF01 + TO Placebo (N=3) | Cohort D2 15 mcg IM CTH522-CAF01 + ID Placebo + TO CTH522 (N=9) | Cohort E1 85 mcg IM CTH522-CAF09b + TO Placebo (N=3) | Cohort E2 85 mcg IM CTH522-CAF09b + ID Placebo + TO CTH522 (N=9) | Cohort F1 IM Placebo + TO Placebo (N=3) | Cohort F2 IM Placebo + ID Placebo + TO Placebo (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 3 (3) | 1 (1) | 3 (3) | 1 (2) | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 1 (3) | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 (2) | 0 | 1 (1) | 0 | 1 (1) | 0 | 1 (1) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Deafness bilateral (Ear and labyrinth disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 2 (2) | 0 | 0
Eye irritation (Eye disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 2 (3) | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 1 (1) | 0
Eyelid irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 (1) | 0 | 3 (4) | 0 | 1 (1) | 1 (3) | 1 (1) | 0 | 0 | 2 (2) | 1 (1)
Ocular discomfort (Eye disorders) | 0 | 2 (3) | 0 | 3 (5) | 0 | 1 (1) | 1 (3) | 0 | 0 | 3 (3) | 2 (3) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 2 (3) | 0 | 1 (1) | 1 (2) | 1 (1) | 0 | 2 (2) | 1 (3) | 0
Swelling of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (2) | 0 | 1 (1) | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2) | 1 (1) | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Nausea (Gastrointestinal disorders) | 0 | 1 (1) | 1 (1) | 0 | 0 | 2 (3) | 1 (1) | 0 | 1 (1) | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 0 | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 | 1 (3) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 2 (2) | 1 (1) | 3 (3) | 1 (2) | 2 (2) | 1 (1) | 4 (5) | 1 (1) | 3 (3) | 0 | 0
Fatigue (General disorders) | 2 (6) | 3 (5) | 1 (1) | 0 | 0 | 4 (7) | 2 (3) | 2 (2) | 0 | 1 (1) | 1 (1) | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 1 (1) | 0 | 2 (2) | 3 (7) | 8 (11) | 0 | 1 (1) | 1 (2) | 4 (6) | 1 (1) | 1 (1)
Injection site movement impairment (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 2 (9) | 9 (37) | 3 (13) | 9 (48) | 3 (11) | 9 (48) | 3 (10) | 9 (42) | 3 (16) | 9 (45) | 2 (4) | 2 (3)
Injection site paraesthesia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 1 (1) | 0 | 2 (2) | 2 (5) | 5 (6) | 0 | 2 (2) | 0 | 2 (3) | 0 | 0
Injection site rash (General disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Injection site swelling (General disorders) | 0 | 1 (2) | 1 (1) | 0 | 2 (4) | 3 (4) | 1 (2) | 1 (1) | 0 | 4 (9) | 0 | 1 (1)
Injection site warmth (General disorders) | 0 | 4 (6) | 2 (4) | 4 (7) | 1 (2) | 6 (11) | 0 | 4 (6) | 1 (1) | 5 (6) | 2 (2) | 1 (3)
Malaise (General disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 0
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gallbladder polyp (Hepatobiliary disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Campylobacter infection (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (1)
Corona virus infection (Infections and infestations) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (1) | 0 | 1 (1)
Gonorrhoea (Infections and infestations) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (2) | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 1 (1)
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Rhinitis (Infections and infestations) | 0 | 2 (3) | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 3 (3) | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (2) | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 (2) | 0 | 1 (1) | 0 | 1 (1) | 0 | 0 | 1 (1) | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 (2) | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Heat stroke (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 (1) | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Mean cell volume decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 2 (2) | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (5) | 1 (1) | 2 (4) | 2 (4) | 3 (4) | 1 (4) | 2 (2) | 2 (3) | 2 (2) | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Pubic pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Anosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (2) | 0 | 1 (1) | 0
Headache (Nervous system disorders) | 0 | 4 (9) | 2 (2) | 4 (4) | 1 (3) | 6 (9) | 1 (4) | 3 (5) | 1 (1) | 2 (6) | 1 (3) | 2 (4)
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 (3) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (2) | 1 (1) | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 | 3 (4) | 1 (1) | 2 (2) | 0 | 0 | 1 (3) | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (4) | 0 | 2 (2) | 0 | 2 (3) | 1 (2) | 1 (1) | 0 | 1 (1) | 2 (3) | 0
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 1 (1) | 2 (2) | 0 | 3 (5) | 1 (1) | 1 (1) | 0 | 1 (1) | 0 | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 | 1 (1) | 0 | 3 (3) | 0 | 2 (3) | 0 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 1 (1) | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 1 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 1 (2) | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0

LIMITATIONS AND CAVEATS:
Screening and recruitment activities had to be paused during the trial due to the Covid-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT03926728/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT03926728/SAP_001.pdf